CLINICAL TRIAL: NCT05115253
Title: Reducing Sedentary Behaviour in Office Workers With a mHealth Health Action Process Approach Intervention and a Just In-Time Adaptive Intervention
Brief Title: Reducing Sedentary Behaviour in Office Workers With a HAPA mHealth Intervention and a Just In-Time Adaptive Intervention
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Western University, Canada (Other)
Responsible Party: Principal Investigator, Dr. Harry Prapavessis, Professor, Western University, Canada
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 119926
Record Dates: First submitted 2021-10-29; First posted 2021-11-10 (Actual); Last update posted 2021-12-23 (Actual); Status verified 2021-12

CONDITIONS: Sedentary Behaviour; Health Behaviour Change
Keywords: Sedentary Behaviour; Health Behaviour Change; HAPA; Health Action Process Approach; JITAI; Just In-Time Adaptive Intervention; Office Workers

STUDY DESIGN:
Intervention Model Description: Upon obtaining consent, eligible participants will be randomly assigned to either of the two intervention groups, a mHealth HAPA group or a JITAI group, or the control group. The study will run for four weeks with the first week acting as a baseline.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- mHealth HAPA Intervention Group (Experimental): This intervention group will receive a single one-on-one online behavioural counselling session and daily personalized SMS text message boosters with the aim of increasing the breaking of consecutive work related sedentary behaviour. Counselling strategies will be grounded in the HAPA model, specifically focusing on the creation of an action plan and the development of coping strategies to increase sedentary behaviour breaks. The SMS text message boosters will be personalized based on participant's preferences of timing, type, frequency, and length. The boosters will framed through HAPA principles with content focusing on risk awareness, outcome expectancy, action and coping planning, barriers and resources, and self-efficacy. The intervention will last for three weeks.
  Interventions: Behavioral: HAPA behavioural counselling + SMS text message boosters
- JITAI Group (Experimental): This intervention group will receive push notifications from a EMA behaviour monitoring mobile application that will be downloaded to each participants' mobile phones. The application will measure and monitor a participant's sedentary behaviour and once a pre-set condition of 30 consecutive sedentary minutes has been reached, the application will administer a push notification notifying the participant to break their sedentary behaviour. The push notifications will ask the participants to stand up, stretch, or lightly walk around to break their current behaviour. The intervention will last for three weeks.
  Interventions: Device: JITAI
- Control Group (No Intervention): The control group will receive no intervention or further instruction past the letter of information.

INTERVENTIONS:
Behavioral: HAPA behavioural counselling + SMS text message boosters — Behavioural counseling grounded in the Health Action Process Approach (HAPA; i.e., action planning and coping planning) paired with daily personalized HAPA guided SMS text message boosters to reduce consecutive workplace sedentary behaviour.
  Arms: mHealth HAPA Intervention Group
Device: JITAI — EMA monitoring mobile phone application that uses a phone's on-board accelerometer to monitor a participant's sedentary behaviour and deliver a push notification once a set condition has been met. This intervention will be utilized to reduce consecutive workplace sedentary behaviour.
  Other Names: mEMA (ilumivu Inc., Boston, MA, www.ilumivu.com)
  Arms: JITAI Group

SUMMARY:
This study will explore the effectiveness of two different interventions, a Health Action Process Approach (HAPA) mobile health (mHealth) intervention and a Just In-Time Adaptive Intervention (JITAI), on reducing sedentary behaviour in office workers. One third of participants will receive the mHealth HAPA intervention, consisting of a theory-driven behavioural counselling session with personalized daily SMS text messages, and another third of participants will receive the JITAI intervention, a behaviour tracking mobile phone application that will alert participants once a set sedentary behaviour condition has been met. The last third of participants will act as a control where they will not receive an intervention or any further information from the letter of information. The study will take place over four weeks, with the first acting as a baseline and the intervention period filling the latter three weeks.

DETAILED DESCRIPTION:
This three-arm repeated measure randomized control trial will randomize participants into two intervention groups and one control group to attempt to reduce sedentary behaviour in office workers. The study will last for four weeks, the first week of the study will be used for baseline measurement and the remaining three weeks used for the intervention.

Participants will be full time office workers primarily recruited from large businesses and corporations. The primary purpose of the study will be to decrease sedentary behaviour in office workers from pre- to post-intervention by breaking up extended periods of sedentary time. The secondary objectives of the study are to compare the effectiveness of each group against one another to assess for any significant differences in sedentary behaviour profiles, total time spent sitting, break frequency, break duration, and time not spent sedentary as well as to examine whether physical activity changed over the course of the intervention.

One intervention group will attempt to reduce sedentary behaviour by receiving push notifications from an EMA tracking mobile phone application after a pre-set sedentary behaviour condition has been met. The application will monitor and collect data from the on-board accelerometer of the participant's phone and when a threshold of 30 consecutive sedentary minutes has been reached, the application will administer a notification asking the participant to break the extended sedentary behaviour they are currently engaged in.

The other intervention group will receive a theory-based behaviour change counselling session paired with daily personalized SMS text message boosters to achieve the study's aims. The counselling sessions and SMS text messages will be framed through the Health Action Process Approach, a behaviour change model that centres around action planning and coping planning. The control group will receive no intervention or further information from the letter of information.

Sedentary behaviour will be collected in the form of duration of time spent sitting, frequency of sedentary behaviour breaks, and duration of sedentary behaviour breaks. These variables will be measured through an EMA tracking mobile phone application that will be downloaded by each participant as well as a weekly online sedentary behaviour questionnaire. Outcome measures will be compared within and between groups to detect differences.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* full-time employee in a desk-based office job (work from home accepted)
* have access to a mobile phone with internet connection
* can read and write in English

Exclusion Criteria:

* any medical or physical limitation that would prevent standing, stretching, and/or light physical activity

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 93 (Estimated)
Dates: Start 2021-12 (Estimated); Primary Completion 2022-03 (Estimated); Study Completion 2022-06 (Estimated)

PRIMARY OUTCOMES:
Changes in Frequency of Breaks from Sitting at Work | Baseline, Weeks 2, 3, 4
  mEMA app (ilumivu Inc., Boston, MA, www.ilumivu.com); accelerometer data Modified version of the SIT-Q 7d (Wijndaele et al., 2014; Sui & Prapavessis, 2016); 1-item; 12-point scale
Changes in Duration of Breaks from Sitting at Work | Baseline, Weeks 2, 3, 4
  mEMA app (ilumivu Inc., Boston, MA, www.ilumivu.com); accelerometer data Modified version of the SIT-Q 7d (Wijndaele et al., 2014; Sui & Prapavessis, 2016); 1-item; 10-point scale
Changes in Time Spent Sitting at Work | Baseline, Weeks 2, 3, 4
  mEMA app (ilumivu Inc., Boston, MA, www.ilumivu.com); accelerometer data Modified version of the SIT-Q 7d (Wijndaele et al., 2014; Sui & Prapavessis, 2016)
Changes in Time Spent Standing at Work | Baseline, Weeks 2, 3, 4
  mEMA app (ilumivu Inc., Boston, MA, www.ilumivu.com); accelerometer data
Changes in Time Spent Engaged in Light Physical Activity at Work | Baseline, Weeks 2, 3, 4
  mEMA app (ilumivu Inc., Boston, MA, www.ilumivu.com); accelerometer data

OTHER OUTCOMES:
Age | Baseline
  Assessed with a single item question: "What is your age?"
Sex | Baseline
  Assessed with a single item question: "What is your sex?"
Gender | Baseline
  Assessed with a single item question: "What gender do you most identify with?"
Ethnicity | Baseline
  Assessed with a single item question: "What ethnicity do you most identify with?"
Height | Baseline
  Assessed with a single item question: "What is your height in either inches or centimetres?"
Weight | Baseline
  Assessed with a single item question: "What is your weight in either pounds or kilograms?"
Work Environment | Baseline
  Assessed with a three item question: "What is your current work environment?"; in office, at home, hybrid
Type of Occupation | Baseline
  Assessed with a four item question: "What general sector does your occupation fall under?"; private, public, charity, other
Hours of Work per Week | Baseline
  Assessed with a single item question: "What are your typical hours of work on an average week?"
Education Level | Baseline
  Assessed with a single item question: "What is your current formal education level?"

CONTACTS AND LOCATIONS:
Overall Officials: Harry Prapavessis, Ph.D, Principal Investigator — Western University
Locations (1):
- The University of Western Ontario, London, Ontario, Canada